CLINICAL TRIAL: NCT04101331
Title: A Phase II Open-label Multicenter Study to Assess the Efficacy and Safety of AFM13 in Patients With Relapsed or Refractory CD30-positive Peripheral T-cell Lymphoma or Transformed Mycosis Fungoides (REDIRECT)
Brief Title: Phase II Study to Assess AFM13 in Patients With R/R CD30-positive T-cell Lymphoma or Transformed Mycosis Fungoides
Acronym: REDIRECT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Affimed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFM13-202
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Peripheral T Cell Lymphoma; Transformed Mycosis Fungoides
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — AFM13

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort A (Experimental): Subjects with Relapsed or Refractory CD30 positive Peripheral T-cell Lymphoma (PTCL).
  Interventions: Drug: AFM13

INTERVENTIONS:
Drug: AFM13 — weekly intravenous infusions of 200mg

SUMMARY:
This is a phase II study to evaluate the antitumor activity and safety of AFM13 given as monotherapy in patients with CD30-positive T-cell lymphoma. The investigational medicinal product AFM13 is a tetravalent bispecific chimeric (anti-human CD30 x anti-human CD16A) recombinant antibody construct which is being developed to treat CD30-positive malignancies.

Patients who suffer from peripheral T-cell lymphoma or transformed mycosis fungoides, whose tumor expresses the surface marker CD30, and who have relapsed after an earlier treatment or have refractory disease will be enrolled into this study if all of the study entry criteria are fulfilled. Dependent on their disease type and the magnitude of CD30 expression, study participants will be assigned to one of 3 study cohorts, each cohort receiving the same treatment of weekly AFM13 infusions (a 200mg dose per infusion).

The main goal of the study is to assess the efficacy of AFM13 treatment as judged by the rate of overall responses. Further goals are to assess the safety of AFM13 treatment, the immunogenicity of AFM13 (as measured by the potential formation of anti-AFM13 antibodies) and the concentration of AFM13 in the blood.

Approx. 1 month after the last dose of AFM13 there will be a final study visit to assess the patients' health status after therapy, followed by quarterly phone contacts to check on their overall health status and long-term survival.

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically confirmed CD30-positive PTCL (most subtypes allowed) or TMF per the revised World Health Organization 2016 classification (Swerdlow, 2016) by central assessment.
* Cohorts A and B (PTCL cohorts): measurable by the modified Lugano Classification (Cheson, 2014); measurable disease of ≥1.5 cm diameter by computed tomography (CT), assessed locally for eligibility. Note: fluorodeoxyglucose (FDG) avid disease by positron emission tomography (PET) recommended, if possible.
* Cohort C (TMF cohort): measurable by the Olsen Criteria (Olsen, 2011) including at least 1 cutaneous lymphoma lesion ≥2 cm in diameter, assessed locally for eligibility.
* Patients must have relapsed or refractory disease AND the following:
* Cohorts A and B (PTCL): patients must have received at least 1 prior line of systemic therapy. For patients with systemic ALCL, patients must have failed or be intolerant to brentuximab vedotin [BV]; Adcetris®
* Cohort C (TMF): patients must have received at least 1 prior line of systemic therapy; and have exhausted systemic therapies with regular approval for their disease

Main Exclusion Criteria:

* Patients with the following subtypes of lymphoma: T-cell prolymphocytic leukemia; T-cell large granular lymphocytic leukemia; Chronic lymphoproliferative disorder of NK cells; Aggressive NK-cell leukemia; Extranodal NK-/T-cell lymphoma; Indolent T-cell lymphoproliferative disorder of the GI tract:
* Has had an allogenic tissue hematopoietic cell/solid organ transplant within the last 3 years. Note: Patients who have had a transplant >3 years ago are eligible as long as there are no signs/symptoms of graft versus host disease (GvHD).
* Requirement for systemic immunosuppressive therapy, e.g. GvHD therapy, <12 weeks prior to the first dose of study drug.
* Prior treatment with AFM13

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2024-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karenza Alexis, MD, Study Director — Affimed Inc.; Won Seog Kim, Dr, Principal Investigator — Samsung Medical Center; Steven Horwitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (69):
- United States (13):
  - University of Alabama at Birmingham (O'Neal Comprehensive Cancer Center), Birmingham, Alabama
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Los Angeles (UCLA) Health, Los Angeles, California
  - Emory University Clinic/Winship Cancer Institute, Atlanta, Georgia
  - Ochsner Clinic Foundation/Precision Cancer Therapies Program, New Orleans, Louisiana
  - University of Michigan Health | Rogel Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Center for Lymphoid Malignancies, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington
- Australia (6):
  - Royal Adelaide Hospital, Adelaide
  - Flinders Medical Centre, Bedford Park
  - Monash Health-Monash Medical Centre, Clayton
  - Concord Repatriation General Hospital, Concord
  - Gosford Hospital, Gosford
  - Linear Clinical Research, Nedlands
- France (5):
  - Centre Hospitalier Universitaire (CHU) de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Brest, Brest
  - CHD Vendée, La Roche-sur-Yon
  - CHU Pontchaillou, Rennes
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Kliniken Essen Sued - Evangelisches Krankenhaus Essen-Werden gGmbH, Essen
  - University Hospital Leipzig, Leipzig
  - Universitaetsmedizin Mainz, Mainz
  - Rotkreuzklinikum Muenchen, München
- Italy (5):
  - Ist.Ematologia E Oncologia Medica L.E A.Seragnoli, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia-Universita degli Studi Di Brescia, Brescia
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST) IRCCS, Meldola
  - Azienda Ospedaliera Niguarda Ca' Granda, Milan
  - Azienda Unita Sanitaria Locale di Ravenna - Ospedale S. Maria delle Croci di Ravenna, Ravenna
- Poland (5):
  - Szpitale Pomorskie Sp. z o.o.. Szpital Morski im. PCK, Oddzial Hematologii i Transplantologii Szpiku, Gdynia
  - Pratia MCM Krakow, Krakow
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie, Klinika Nowotworow Ukladu Chlonnego, Warsaw
  - Instytut Hematologii i Transfuzjologii, Klinika Hematologii, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu. Klinika Hematologii, Nowotworow Krwi i Transplantacji Szpiku, Wroclaw
- Russia (6):
  - Republic Hospital n.a. V.A. Baranov, Petrozavodsk
  - First State Saint-Petersburg Pavlov Medical University, Saint Petersburg
  - GUZ Leningrad Regional Clinical Hospital, Saint Petersburg
  - Russian Research Institute of Hematology and Transfusiology of the Federal Biomedical Agency, Saint Petersburg
  - Saratov State Medical University, Saratov
  - Regional Clinical Hospital, Tula
- South Korea (5):
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (10):
  - Duran I Reynals Hospital Catalan Institute Of Oncology, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia Badalona, Hospital Germans Trias I Pujol, Barcelona
  - Institut Catala d' Oncologia Girona, Girona
  - Hospital Universitario 12 de Octubre-Centro de Actividades Ambulatorias, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Institut Catala d'Oncologia Tarragona, Tarragona
- Turkey (Türkiye) (10):
  - Ankara University Faculty of Medicine, Department of Internal Diseases, Hematology Division, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim Arastirma Hastanesi Hematoloji Klinigi Ankara, Ankara
  - Gazi University Faculty of Medicine, Department of Internal Diseases, Ankara
  - Sağlık Bilimleri Üniversitesi Gülhane Eğitim ve Araştırm Hastanesi, Ankara
  - Istanbul Universitesi Istanbul Tip Fakultesi Ic Hastaliklari Anabilim Dali Hematoloji Bilim Dali Fatih, Istanbul
  - Ege University Medical Faculty, Izmir
  - Kocaeli University Faculty of Medicine, Department of Internal Diseases, Hematology Division, İzmit
  - Ondokuz Mayis Universitesi Tip Fakultesi Saglik Uyg. ve Egitim Merkezi, Samsun
  - Tekirdag Namik Kemal Universitesi Saglik Uygulama ve Arastirma Hastanesi, Tekirdağ
  - KaradenizTeknik Universitesi Tip Fakultesi Farabi Hastanesi, Trabzon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a Phase II open-label multicenter study to assess the efficacy and safety of AFM13 in subjects with relapsed or refractory CD30-positive peripheral T-cell lymphoma.
Pre-assignment Details: All the subjects were screened for CD30 expression. Investigators assessed the subjects, and they were enrolled in the study if they met all inclusion criteria and none of the exclusion criteria.
Period: Overall Study
Arm/Group | Cohort A
Started | 108
Completed | 3
Not Completed | 105
Not completed — Adverse Event | 9
Not completed — Disease progression | 82
Not completed — Withdrawal by Subject | 1
Not completed — Investigator decision | 6
Not completed — Death | 6
Not completed — Allogenic transplant | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): consist of all subjects who received at least one dose of AFM13.
Arm/Group | Cohort A
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (13.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 90
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 75
  More than one race | 0
  Unknown or Not Reported | 13

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Assessed by Independent Review Committee Based on PET-CT
Description: Overall response by Positron Emission Tomography-Computed Tomography (PET-CT) as defined by achieving complete response and/or partial response assessed by an Independent Review Committee (IRC) utilizing the modified Lugano Classification Revised Staging System for malignant lymphoma (Cheson, 2014).
Time Frame: Tumor assessment performed every 8 weeks for first 3 assessments, then every 12 weeks until documented disease progression (up to 28 months).
Population: The full analysis set (FAS) followed the intent to treat (ITT) principle and consisted of all subjects who received at least one dose of AFM13.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Cohort A
Number analyzed (Participants) | 108
percentage | 32.4 [23.7 to 42.1]
Statistical Analysis 1: Comparison: Cohort A; Test type: Other; p = 0.051, Exact binomial test — One-sided p-value; Exact binomial test compares versus a proportion of 0.25

2. Secondary Outcome: Overall Response Rate Assessed by Investigator Based on PET-CT
Description: Overall response by Positron Emission Tomography-Computed Tomography (PET-CT) as defined by achieving complete response and/or partial response assessed by the investigator utilizing the modified Lugano Classification Revised Staging System for malignant lymphoma (Cheson, 2014).
Time Frame: Tumor assessment performed every 8 weeks for first 3 assessments, then every 12 weeks until documented disease progression (up to 46 months).
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Cohort A
Number analyzed (Participants) | 108
percentage | 32.4 [23.7 to 42.1]
Statistical Analysis 1: Comparison: Cohort A; Test type: Other; p = 0.051, Exact binomial test — One-sided p-value; Exact binomial test compares versus a proportion of 0.25

3. Secondary Outcome: Overall Response Rate Assessed by Investigator Based on CT
Description: Overall response by Computed Tomography (CT) as defined by achieving complete response and/or partial response assessed by the investigator utilizing the modified Lugano Classification Revised Staging System for malignant lymphoma (Cheson, 2014).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Cohort A
Number analyzed (Participants) | 108
percentage | 30.6 [22.1 to 40.2]
Statistical Analysis 1: Comparison: Cohort A; Test type: Other; p = 0.112, Exact binomial test — One-sided p-value; Exact binomial test compares versus a proportion of 0.25

4. Secondary Outcome: Complete Response Rate and Partial Response Rate Assessed by Independent Review Committee Based on PET-CT
Description: Complete response and/or partial response by Positron Emission Tomography-Computed Tomography (PET-CT) assessed by an Independent Review Committee (IRC) utilizing the modified Lugano Classification Revised Staging System for malignant lymphoma (Cheson, 2014).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Cohort A
Number analyzed (Participants) | 108
percentage
  Complete response rate (CR rate) | 12.0 [6.6 to 19.7]
  Partial response rate (PR rate) | 20.4 [13.2 to 29.2]

5. Secondary Outcome: Complete Response Rate, Partial Response Rate and Overall Response Rate Assessed by Independent Review Committee Based on CT
Description: Overall response by Computed Tomography (CT) as defined by achieving complete response and/or partial response assessed by an Independent Review Committee (IRC) utilizing the modified Lugano Classification Revised Staging System for malignant lymphoma (Cheson, 2014).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Cohort A
Number analyzed (Participants) | 108
percentage
  Overall response rate (ORR) | 25.0 [17.2 to 34.3]
  Complete response rate (CR rate) | 7.4 [3.3 to 14.1]
  Partial response rate (PR rate) | 17.6 [10.9 to 26.1]
Statistical Analysis 1: Comparison: Cohort A; Test type: Other; p = 0.537, Exact binomial test — One-sided p-value; Exact binomial test compares versus a proportion of 0.25

6. Secondary Outcome: Duration of Overall Response Assessed by Independent Review Committee Based on PET-CT
Description: Duration of response (DOR) defined as the period from first Partial Response (PR) and Complete Response (CR) assessment till first assessment of progressive disease or death. Response assessed by Positron Emission Tomography-Computed Tomography (PET-CT) by Independent Review Committee (IRC).
Time Frame: as for outcome 2
Population: All subjects of the full analysis set (FAS) who had a response in PET assessed by IRC.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A
Number analyzed (Participants) | 35
months | 2.3 [1.9 to 8.7]

7. Secondary Outcome: Duration of Overall Response Assessed by Independent Review Committee Based on CT
Description: Duration of response (DOR) defined as the period from first Partial Response (PR) and Complete Response (CR) assessment till first assessment of progressive disease or death. Response assessed by Computed Tomography (CT) by Independent Review Committee (IRC).
Time Frame: as for outcome 2
Population: All subjects of the full analysis set (FAS) who had a response in CT assessed by IRC.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A
Number analyzed (Participants) | 27
months | 5.3 [1.9 to 6.9]

8. Secondary Outcome: Duration of Overall Response Assessed by Investigator Based on PET-CT
Description: Duration of response (DOR) defined as the period from first Partial Response (PR) and Complete Response (CR) assessment till first assessment of progressive disease or death. Response assessed by Positron Emission Tomography-Computed Tomography (PET-CT) by the investigator.
Time Frame: as for outcome 2
Population: All subjects of the full analysis set (FAS) who had a response in PET-CT assessed by investigator.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A
Number analyzed (Participants) | 35
months | 3.3 [1.9 to 8.7]

9. Secondary Outcome: Duration of Overall Response Assessed by Investigator Based on CT
Description: Duration of response (DOR) defined as the period from first Partial Response (PR) and Complete Response (CR) assessment till first assessment of progressive disease or death. Response assessed by Computed Tomography (CT) by the investigator.
Time Frame: as for outcome 2
Population: All subjects of the full analysis set (FAS) who had a response in CT assessed by investigator.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A
Number analyzed (Participants) | 33
months | 6.3 [2.0 to 8.7]

10. Secondary Outcome: Number of Subjects With Treatment Related Adverse Event
Description: Number of subjects who had treatment (AFM13) related Adverse Events.
Time Frame: From the date of first treatment until the date of the last treatment + 37 days, up to 199 weeks.
Population: The safety set consisted of all subjects who received at least one dose of AFM13 and had at least one post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A
Number analyzed (Participants) | 108
Participants | 105

11. Secondary Outcome: Maximum Measured Concentration (Cmax) of AFM13
Description: Maximum measured concentration (Cmax) of the AFM13 in serum. Geometric coefficient of variation is given in percentages.
Time Frame: Predose and 1 hour after start of infusion, end of injection (EOI) and 1 hour, 2 hours, 3 hours, 24 hours and 48 hours after EOI on Cycle 1 Day 1 and Day 29.
Population: The pharmacokinetic set (PK) consists of subjects who had at least received one dose of study drug and had at least one post dose PK measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Cohort A
Number analyzed (Participants) | 20
Nanogram/milliliter
  Cycle 1 - day 1 | 26232 (270)
  Cycle 1 - day 29: number analyzed (Participants) | 16
  Cycle 1 - day 29 | 24435 (364)

12. Secondary Outcome: Area Under the Concentration-Time Curve of AFM13 From 0 to Infinity (AUC 0-∞)
Description: Area under concentration (AUC) versus time curve of the AFM13 in serum over time interval from 0 extrapolated to infinity.
  Geometric coefficient of variation is given in percentages.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter
Arm/Group | Cohort A
Number analyzed (Participants) | 18
nanogram*hour/milliliter
  Cycle 1 - day 1 | 612361 (60.3)
  Cycle 1 - day 29: number analyzed (Participants) | 13
  Cycle 1 - day 29 | 749717 (35)

13. Secondary Outcome: Volume of Distribution at Steady State (Vss) of AFM13
Description: Volume of distribution at steady state (Vss) of the AFM13. Geometric coefficient of variation is given in percentages.
Time Frame: Predose and 1 hour after start of infusion, end of injection (EOI) and 1 hour, 2 hours, 3 hours, 24 hours and 48 hours after EOI on Cycle 1 Day 29.
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Cohort A
Number analyzed (Participants) | 13
Liter | 5.1 (58.4)

14. Secondary Outcome: The Terminal Half-life (t1/2) of AFM13
Description: The terminal half-life (t1/2) of the AFM13. Geometric coefficient of variation is given in percentages.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Cohort A
Number analyzed (Participants) | 18
hour
  Cycle 1 - day 1 | 20.7 (35.9)
  Cycle 1 - day 29: number analyzed (Participants) | 13
  Cycle 1 - day 29 | 19.6 (47.4)

15. Secondary Outcome: European Quality of Life 5-dimensional Pain/Discomfort Score (EQ-5D)
Description: Quality of Life (QoL) as measured by the European QoL 5-dimensional questionnaire (EQ-5D) for Cohorts A. The EQ-5D comprises asks for the current health state in the five dimensions: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Pain/discomfort scores assessed based on questionnaire. The categories of the response offer three levels pain/discomfort score: "no pain or discomfort" (score of 1), "moderate pain or discomfort" (score of 2), and "extreme pain and discomfort" (score of 3). Scores are presented from baseline to each visit for Cohort A.
Time Frame: At baseline and final study visit, up to 199 weeks.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A
Number analyzed (Participants) | 108
Participants
  Baseline: No pain or discomfort | 41
  Baseline: Moderate pain or discomfort | 55
  Baseline: Extreme pain or discomfort | 9
  Baseline: Missing | 3
  Final Study Visit: No pain or discomfort | 19
  Final Study Visit: Moderate pain or discomfort | 38
  Final Study Visit: Extreme pain or discomfort | 5
  Final Study Visit: Missing | 46

16. Secondary Outcome: European Quality of Life 5-dimensional Visual Analogue Scale Scores (EQ-5D)
Description: Quality of Life (QoL) as measured by the European Quality of Life 5-dimensional questionnaire (EQ-5D) for Cohorts A. Visual Analogue Scale scores assessed based on drawn scale from 0(worst imaginable state) to 100(best imaginable state). Subjects chose their health state on scale based on their situation by themselves. A negative outcome indicates a decrease in score compared to the baseline value.
Time Frame: From baseline until final study visit, up to 199 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A
Number analyzed (Participants) | 108
score on a scale | -9.16 (25.46)

17. Secondary Outcome: Number of Subjects Who Developed Anti-drug Antibodies (ADA) During Treatment
Description: Number of subjects who had treatment (AFM13) and developed anti-drug antibodies (ADA).
Time Frame: Pre-dose Day 1 on cycle 1 and end of treatment, up to approximately 46 months.
Population: The safety set consisted of all subjects who received at least one dose of AFM13and had at least one post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A
Number analyzed (Participants) | 108
Participants | 21

ADVERSE EVENTS:
Time Frame: From the date of first treatment till the date of the last treatment + 37 days, up to 199 weeks.
Description: The safety set consisted of all subjects who received at least one dose of AFM13 and had at least one post-baseline safety assessment.
Arm/Group | Cohort A
All-Cause Mortality (participants affected / at risk) | 52/108
Serious Adverse Events (participants affected / at risk) | 44/108
Other Adverse Events (participants affected / at risk) | 95/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=108)
COVID-19 (Infections and infestations) | 9
Pneumonia (Infections and infestations) | 6
Herpes zoster (Infections and infestations) | 2
Septic shock (Infections and infestations) | 2
COVID-19 pneumonia (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 1
Enterococcal bacteraemia (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Pneumonia aspiration (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Rhinovirus infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Streptococcal bacteraemia (Infections and infestations) | 1
Vascular access site infection (Infections and infestations) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 5
Pyrexia (General disorders) | 2
Chills (General disorders) | 1
General physical health deterioration (General disorders) | 1
Pain (General disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Acute left ventricular failure (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Hepatic enzyme increased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1
Bronchitis (Infections and infestations) | 1
Device Related Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=108)
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 17
Erythema (Skin and subcutaneous tissue disorders) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 7
Anaemia (Blood and lymphatic system disorders) | 16
Neutropenia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Lymphopenia (Blood and lymphatic system disorders) | 7
Pyrexia (General disorders) | 21
Asthenia (General disorders) | 9
Chills (General disorders) | 7
Infusion related reaction (Injury, poisoning and procedural complications) | 25
Hypokalaemia (Metabolism and nutrition disorders) | 9
Decreased appetite (Metabolism and nutrition disorders) | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Headache (Nervous system disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Insomnia (Psychiatric disorders) | 8
Upper respiratory tract infection (Infections and infestations) | 6
Blood lactate dehydrogenase increased (Investigations) | 6
Respiratory Tract Infection (Infections and infestations) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor has the right to review communications for 90 days prior to public release (whereby the sponsor may ask to consider modifications to ensure necessary protection of sponsor's IP). Any publication shall be not made before the first multi-centre publication if the study is a part of a multi-centred clinical trial. Also, if a publication concerns the analyses of data from a multi-centred clinical trial, the communication shall make reference to the relevant multi-centre publication

DOCUMENTS (2):
  • Study Protocol (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/31/NCT04101331/Prot_002.pdf
  • Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/31/NCT04101331/SAP_001.pdf